CLINICAL TRIAL: NCT04798924
Title: Visual Rehabilitation After Occipital Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Krystel Huxlin, James V. Aquavella Professor of Ophthalmology, Associate Chair for Research, Dept. Ophthalmology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00005966; R01EY027314 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Stroke, Ischemic; Quadrantanopia; Vision Loss Partial; Visual Field Defect, Peripheral; Peripheral Visual Field Defect of Both Eyes; Peripheral Visual Field Defect; Hemianopsia; Hemianopia; Homonymous Hemianopia; Homonymous Hemianopsia; Visual Fields Hemianopsia; Occipital Lobe Infarct; Quadrantanopsia; Stroke Hemorrhagic
Keywords: Occipital stroke; vision loss; Homonymous quadrantanopia; Homonymous quadrantanopsia; stroke; Vision loss after stroke; Vision recovery; Vision restoration; Partial vision loss
MeSH Terms: conditions — Ischemic Stroke; Hemianopsia; Hemorrhagic Stroke; Vision Disorders; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Training in the blind field (Experimental): Training in the blind field using specialized software
  Interventions: Device: Subacute Training in the blind field; Device: Chronic Training in the blind field
- Training in the intact field (Experimental): Training in the intact field using specialized software
  Interventions: Device: Subacute Training in the intact field; Device: Chronic Training in the blind field

INTERVENTIONS:
Device: Subacute Training in the intact field — A computer software and chin-rest necessary to perform visual training will be loaned to each subject to be used at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a predetermined location in the intact field. The computer program will automatically create a record of patient performance during each home training session. Subjects will train daily (about 40-60 minutes total), 5 to 7 days per week for at least one and up to 6 months.
  Arms: Training in the intact field
Device: Subacute Training in the blind field — A computer software and chin-rest necessary to perform visual training will be loaned to each subject to be used at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a predetermined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. Subjects will train daily (about 40-60 minutes total), 5 to 7 days per week for at least one and up to 6 months.
  Arms: Training in the blind field
Device: Chronic Training in the blind field — After the initial training period of one to six months, the same computer software will continue to be used for all subjects. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a predetermined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. Subjects will train daily (about 40-60 minutes total), 5 to 7 days per week for at least 6 months.

SUMMARY:
This research aims to examine changes in plastic potential of the visual system with time from stroke affecting primary visual cortex. We will measure structural and mechanistic aspects of progressive degeneration along the early visual pathways, correlating them with changes in visual performance, and in responsiveness to visual restoration training. This project will advance both scientific knowledge, as well as technical capability and clinical practices for restoring vision and quality of life for people suffering from cortical blindness.

ELIGIBILITY:
Inclusion Criteria:

* Residents of US and Canada
* MRI and/or CT scans showing evidence of one-sided / unilateral stroke or stroke-like damage to the primary visual cortex or its immediate afferent white matter sustained less than 6-months prior to enrollment
* Reliable visual field defects in both eyes as measured by Humphrey, Macular Integrity Assessment (MAIA), Goldmann, and/or equivalent perimetry. This deficit must be large enough to enclose a 5-deg diameter visual stimulus.
* Ability to fixate on visual targets reliably for 1000ms (as demonstrated by visual fields, and verified in study participation)
* Willing and safely able to undergo magnetic resonance imaging (MRI) scanning
* Willing, able, and competent to provide informed consent
* Fluent in written and spoken English
* Cognitively able, responsible, and willing to complete daily visual training independently at home for several months.

Exclusion Criteria:

* Past or present ocular disease interfering with vision
* Best corrected visual acuity worse than 20/40 in either eye
* Presence of damage to the dorsal Lateral Geniculate Nucleus, as shown on MRI/CT scans
* Diffuse, whole brain degenerative processes
* Brain damage deemed by study staff to potentially interfere with training ability or outcome measures
* History of traumatic brain injury
* Documented history of drug/alcohol abuse
* Currently use of neuroactive medications which would impact training, as determined by PI
* Cognitive or seizure disorders
* One-sided attentional neglect
* Inability to perform the visual training exercises as directed

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Direction Discrimination Threshold | baseline, 6 months, 12 months
  For each subject, we will measure the ability to detect differences in the motion direction of visual stimuli relative to horizontal, measured in degrees of visual angle. These assessments will be based on what can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline to 6-months post-stroke, then 6- to 12-months post stroke, and baseline to 12-months.**
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.

SECONDARY OUTCOMES:
Direction Integration Threshold | baseline, 6 months, 12 months
  This will measure the ability of subjects to integrate across a range of motion directions measured in degrees of visual angle. These assessments will be based on what range of motion directions can be reliably integrated at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline to 6-months post-stroke, then 6- to 12-months post stroke, and baseline to 12-months.
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Contrast Sensitivity for Direction | baseline, 6 months, 12 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for direction discrimination.
  For each subject, we will measure the ability to correctly detect the motion direction of visual stimuli that are also varying in contrast against a grey background. We will measure the luminance contrast that can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline to 6-months post-stroke, then 6- to 12-months post stroke, and baseline to 12-months.
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
contrast sensitivity for static orientation | baseline, 6 months, 12 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for static orientation discrimination.
  For each subject, we will measure the ability to correctly detect the orientation of non-moving visual stimuli that vary in contrast against a grey background. We will measure the luminance that can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline to 6-months post-stroke, then 6- to 12-months post stroke, and baseline to 12-months.
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Ganglion cell complex thickness laterality | baseline, 6 months, 12 months
  Change in thickness of the ganglion cell complex will be measured by retinal optical coherence tomography (OCT) scans from baseline to 6- and 12- months post stroke.**
  We will perform OCT imaging of the foveal region of the retina (6mm ETDRS) in both eyes of each patient. Images will be automatically segmented. Estimated thickness of the ganglion cell complex will be extracted and aligned with estimates of the blind field's visual sensitivity obtained from fundus-controlled MAIA perimetry. We will then compute a laterality index LI as follows: LIGCCT=(Tc-Ti)/(Tc+Ti) where Tc=thickness in the control lateral OCT quadrant, Ti=thickness in the impaired lateral OCT quadrant.
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Ganglion cell complex volume laterality | baseline, 6 months, 12 months
  Change in volume of the ganglion cell complex will be measured by retinal optical coherence tomography (OCT) scans from baseline to 6- and 12- months post stroke.**
  We will perform OCT imaging of the foveal region of the retina (6mm ETDRS) in both eyes of each patient. Images will be automatically segmented. Estimated volume of the ganglion cell complex will be extracted and aligned with estimates of the blind field's visual sensitivity obtained from fundus-controlled MAIA perimetry. We will then compute a laterality index as follows: LIGCCT=(Tc-Ti)/(Tc+Ti) where Tc=thickness in the control lateral OCT quadrant, Ti=thickness in the impaired lateral OCT quadrant.
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Optic Tract (OT) laterality | baseline, 6 months, 12 months
  OT volume analysis will be performed from high resolution structural T1 MRI images of the brain. Mirrored masks of equal size will be hand-drawn over the OTs in each brain slice of a given subject, starting three slices posterior to the optic chiasm and continuing posteriorly until the OTs are no longer distinct from surrounding structures. The volume of each optic tract will be calculated from these masks by first establishing the maximum voxel intensity (range from 0 to 255) across the two OTs, then counting the number of voxels in each OT mask with brightness values between 5 and 85% of this maximum. We will then compute an OT laterality Index (LI85) to represent the relative difference in estimated volume between the two OTs of each participant, where LI85=(OTc-OTi)/(OTc+OTi), where OTc=number of voxels with brightness 5-85% of maximum in the contralesional OT and OTi = number of voxels with brightness 5-85% of maximum in the ipsilesional OT.

OTHER OUTCOMES:
MAIA Visual Field Perimetry | baseline, 6 months, 12 months
  We will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system. These changes will be measured and compared between baseline, 6-months post stroke, and 12 months post stroke.**
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Humphrey 10-2 and 24-2 perimetry | baseline, 6 months, 12 months
  We will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system. These changes will be measured and compared between baseline, 6-months post stroke, and 12 months post stroke.**
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.
Goldmann perimetry | baseline, 6 months, 12 months
  We will measure the change in area of vision (degrees squared) as encompassed by each isopter, measured by one of 3 different light stimuli.
  The 3 isopters we will compare are:
  1. I2e 1asb, 0.25 mm^2
  2. I4e 10asb, 0.25 mm^2
  3. V4e 1000asb, 64 mm^2
  These changes will be measured and compared between baseline, 6-months post stroke, and 12 months post stroke.**
  **NOTE: Our protocol allows for a +1 month variance for all timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States